CLINICAL TRIAL: NCT01328522
Title: Comparison of the Safety and Pharmacokinetics of Two SAR153191 (REGN88) Drug Products in Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PKM12058; U1111-1119-2883 (Other: UTN)
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAR153191 drug product 1 (Experimental): SAR153191 drug product 1 in a single injection.
  Methotrexate (stable dose) and folic/folinic acid are continued as background therapy.
  Interventions: Drug: SAR153191 (REGN88)
- SAR153191 drug product 2 (Experimental): SAR153191 drug product 2 in a single injection.
  Methotrexate (stable dose) and folic/folinic acid are continued as background therapy.
  Interventions: Drug: SAR153191 (REGN88)

INTERVENTIONS:
Drug: SAR153191 (REGN88) — Pharmaceutical form:solution
  Route of administration: subcutaneous

SUMMARY:
Primary Objective:

Assess the comparative safety and tolerability of two SAR153191 (REGN88) drug products after a single dose administration in rheumatoid arthritis patients.

Secondary Objective:

Assess the comparative pharmacokinetic profiles of the two SAR153191 (REGN88) drug products after a single dose administration in rheumatoid arthritis patients.

DETAILED DESCRIPTION:
The duration of the study period per subject is 5-7 weeks broken down as follows:

* Screening: 1 to 14 days,
* Treatment: 1 day (2 overnight stays at the study site),
* Follow-up: up to 5 weeks after dosing (an additional outpatient follow-up may be scheduled depending on the last results).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of rheumatoid arthritis (RA) > or = 3 months duration.
* Treated for a minimum of 12 weeks with Methotrexate (MTX) prior to randomization. Treatment must be continued on a stable dose for the duration of the study.

Exclusion criteria:

* Autoimmune disease other than RA.
* History of acute inflammatory joint disease other than RA.
* Surgery within 4 weeks prior to the screening visit or with planned elective surgery within the next 3 months.
* Latent or active tuberculosis.
* Fever (≥38 C) or persistent chronic or active recurring infection requiring treatment with antibiotics, antivirals, or antifungals within 4 weeks prior to the screening visit, or history of frequent recurrent infections.
* Received administration of any live (attenuated) vaccine within 3 months prior to the randomization visit (eg, varicella-zoster vaccine, oral polio, rabies).
* Received tuberculosis vaccination within 12 months prior to screening
* Prior therapy with a Tumor Necrosis Factor (TNF) antagonist or any other biologic agents within 3 months prior to inclusion.
* Known latex sensitivity.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of potentially clinically significant abnormalities in clinical laboratory test results | 5 weeks
Occurrence of Adverse Events | 5 weeks

SECONDARY OUTCOMES:
Pain evaluation using the Present Pain Intensity (PPI) verbal questionnaire | 2 days
Pain evaluation using Visual Analog Scale (VAS) | 2 days
Diameter of the erythema at injection site | 2 days
Diameter of the edema at injection site | 2 days
Serum concentration of SAR153191: Maximum plasma concentration (Cmax), first time to reach Cmax (tmax), area under the plasma concentration (AUClast and AUC) | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- United States (4):
  - Investigational Site Number 840003, Beverly Hills, California
  - Investigational Site Number 840001, Ocala, Florida
  - Investigational Site Number 840004, Duncansville, Pennsylvania
  - Investigational Site Number 840002, Dallas, Texas